CLINICAL TRIAL: NCT06156072
Title: Use of Ultrasound for Blood Sample Drawing for Microbiological Analysis in Critically Ill Patients:he ECOVEN Feasibility Study
Brief Title: Ultrasound-guided Blood Sampling Drawing for Microbiological Analysis in the Critically Ill
Acronym: ECOVEN
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, LA BELLA MARIACARMEN, Nurse, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 6046
Record Dates: First submitted 2023-11-21; First posted 2023-12-05 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Sepsis; Septic Shock; Infections; Diagnosis
MeSH Terms: conditions — Sepsis; Shock, Septic; Infections; Disease

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patient requiring blood culture: After the request of treating physician of blood culture, each patient deemed eligible, will undergo the prescirbed couple of peripheral blood samples. The first one will be done with the classical blind technique, while the second one with ultrasound guidance.
  Interventions: Diagnostic Test: Ultrasound-guided venipuncture

INTERVENTIONS:
Diagnostic Test: Ultrasound-guided venipuncture — Venipuncture will be performed using ultrasound to identify the most appropriate vessel and guide the puncture

SUMMARY:
This study will test the feasibility of ultrasound-guided sterile blood sampling for critically ill patients with suspected sepsis requiring blood culture. The aim of the study is to evaluate the feasibility and safety of the use of ultrasound for blood cultures in a population of patients which can present difficult venous access and requiring more than one venipuncture attempt in general clinical practice

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 year-old)
* admitted to intensive care unit
* suspected sepsis requiring blood cultrure

Exclusion Criteria:

* pregnancy
* infections requiring respiratory isolation
* burns or skin disease involving arms and/or more than 60% of body surface

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Alla adult patients admitted to ICU with a suspected sepsis will be enrolled, when treating physician will prescribe blood culture for microbiological analysis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of attempted venipunctures | One hour after clinical decision of blood culture execution
  Evaluation of the feasibility of ultrasound-guided venipuncture for blood samples in patients requiring ,microbiological analysis. Feasibility will be evaluated in terms of number of needed attempts of venipuncture

SECONDARY OUTCOMES:
Incidence of possible complications (accidental arterial puncture, visible ematoma) | One hour after clinical decision of blood culture execution
  Evaluation of safety of venipuncture in terms of possible complications (accidental arterial puncture, ematoma)
Incidence of contamination of ultrasound-guided venipuncture | One hour after clinical decision of blood culture execution
  Evaluation of blood sample bacterial contamination compared to blind puncture

CONTACTS AND LOCATIONS:
Overall Officials: Antonio M Dell'Anna, M.D., Study Chair — Fondazione Policlinico Universitario A. Gemelli, IRCCS

IPD SHARING:
Plan to Share IPD: Undecided